CLINICAL TRIAL: NCT00449033
Title: A Phase III Randomized, Double-blind, Placebo Controlled Trial Comparing the Efficacy of Gemcitabine, Cisplatin and Sorafenib to Gemcitabine, Cisplatin and Placebo in First-Line Treatment of Patients With Stage IIIb With Effusion and Stage IV Non-Small Cell Lung Cancer (NSCLC)
Acronym: NEXUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12006; 2006-002688-26 (EudraCT Number)
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Results first posted 2011-09-09 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small Cell Lung Cancer (NSCLC); Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Sorafenib; Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib (Nexavar, BAY43-9006) + GC (Experimental): Up to 6 cycles (21 days per cycle) of gemcitabine (G) and cisplatin (C) with sorafenib. Day 1: gemcitabine 1250 mg/ m^2 infusion (IV), followed by cisplatin 75 mg/ m^2 IV; Day 8: gemcitabine 1250 mg/ m^2 IV; Days 1-21: sorafenib 2 tablets (200 mg) taken orally (po) twice daily (bid). If the patient had radiological evidence of stable disease (SD) or better after completing up to 6 cycles in the Chemotherapy Phase, the patient could continue to Maintenance Phase, during which sorafenib was administered 400 mg bid until criteria for withdrawal were met.
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006); Drug: Gemcitabine; Drug: Cisplatin
- Placebo + GC (Placebo Comparator): Up to 6 cycles (21 days per cycle) of gemcitabine (G) and cisplatin (C) with placebo. Day 1: gemcitabine 1250 mg/ m^2 infusion (IV), followed by cisplatin 75 mg/ m^2 IV; Day 8: gemcitabine 1250 mg/ m^2 IV; Days 1-21: placebo 2 tablets po bid. If the patient had radiological evidence of SD or better after completing up to 6 cycles in the Chemotherapy Phase, the patient could continue to Maintenance Phase, during which 2 placebo tablets were administered bid until criteria for withdrawal were met.
  Interventions: Drug: Placebo; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Multikinase inhibitor, Sorafenib 400 mg po bid; applied in combination with chemotherapy components: Gemcitabine 1250 mg/m^2 IV, Cisplatin 75 mg/m^2 IV
  Arms: Sorafenib (Nexavar, BAY43-9006) + GC
Drug: Placebo — Placebo 2 tablets po bid; applied in combination with chemotherapy components: Gemcitabine 1250 mg/m^2 IV, Cisplatin 75 mg/m^2 IV
  Arms: Placebo + GC
Drug: Gemcitabine — Chemotherapy component; Gemcitabine 1250 mg/m^2 IV
Drug: Cisplatin — Chemotherapy component; Cisplatin 75 mg/m^2 IV

SUMMARY:
Evaluation of gemcitabine and cisplatin in combination with either sorafenib or placebo for the treatment of patients with advanced Non-Small Cell Lung Cancer (NSCLC)

DETAILED DESCRIPTION:
During follow-up, it was determined that there was one additional patient on placebo that was still receiving treatment as of 06 APR 2010 and therefore 10 patients' data are reported in the current CSR addendum, 6 in the sorafenib + GC group and 4 in the placebo + GC group, and as before all in the ITT (non-squamous) population.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Stage IIIB (with cytologically confirmed malignant pleural or pericardial effusion) or Stage IV histological or cytological confirmation of NSCLC of non-squamous cell carcinoma subtype. (thoracentesis or pericardiocentesis is not necessary if a biopsy of the original tumor is available to confirm diagnosis of NSCLC).
* Patients with at least one measurable lesion. Lesions must be measured by CT-scan or MRI (Magnetic resonance imaging) according to Response Evaluation Criteria in Solid Tumors (RECIST, see Appendix 10.3)
* Life expectancy of at least 12 weeks
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to start of first dose:
* Hemoglobin >/= 9.0 g/dl (>/= 5.6 mmol/l)
* Absolute neutrophil count (ANC) >/= 1,500/mm3
* Platelet count >/= 100,000/µl
* Total bilirubin </= 1.5 x upper limit of normal
* Alanine transaminase (ALT) and Aspartate transaminase (AST) </= 2.5 x upper limit of normal (</= 5 x upper limit of normal for patients with liver involvement of their cancer)
* Alkaline Phosphatase </= 4 x upper limit of normal
* PT-INR (Prothrombin Time - International Normalized Ratio) (international normalized ratio of PT) /PTT (Partial Thromboplastin Time) < 1.5 x upper limit of normal
* Serum Creatinine </= 1.5 times the upper limit of normal and Serum Creatinine Clearance >/= 70ml/min
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to performing any study specific procedures.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.

Exclusion Criteria:

* Excluded medical conditions:

  * Cardiac disease: Congestive heart failure > class II NYHA (New York Heart Association). Patients must not have unstable angina (anginal symptoms at rest) or active coronary artery disease (CAD), or myocardial infarction within the past 6 months
  * Cardiac arrhythmias requiring anti-arrhythmic therapy
  * Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
  * History of HIV (Human immunodeficiency virus) infection or chronic hepatitis B or C
  * Active clinically serious infections (> grade 2 NCI-CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) version 3.0)
  * Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
  * Known brain metastasis. Patients with neurological symptoms should undergo a CT scan/MRI of the brain to exclude brain metastasis.
  * History of organ allograft
  * Patients with evidence or history of bleeding diathesis or coagulopathy
  * Patients undergoing renal dialysis
  * Cancer other than NSCLC within 5 years prior to start of study treatment EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, or superficial bladder tumors [Ta (Noninvasive tumor), Tis (Carcinoma in situ) & T1 (Tumor invades lamina propria)]
  * Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
  * Thrombotic or embolic events such as cerebrovascular accident including transient ischemic attacks within the past 6 months
  * Pulmonary hemorrhage/bleeding event > Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 within 4 weeks of first dose of study drug
  * Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
  * Serious, non-healing wound, ulcer, or bone fracture
  * Uncorrected dehydration
  * Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must use adequate birth control measures during the course of the trial. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
  * Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
  * Known or suspected allergy to the investigational agent or any agent given in association with this trial
  * Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
  * Patients unable to swallow oral medications
  * Any malabsorption condition
  * Patients with a hearing impairment (FOR GERMANY ONLY)
  * NSCLC patients with squamous cell carcinoma diagnosis documented either by cytology or biopsy.
* Excluded therapies and medications, previous and concomitant:

  * Any prior systemic anticancer therapy including cytotoxic therapy, targeted agents, experimental therapy, adjuvant, or neo-adjuvant therapy for NSCLC
  * Concomitant use of nephrotoxic drugs, ototoxic drugs, anticonvulsant, anti-gout treatment
  * Radiotherapy during study or within 3 weeks of start of study drug. (Palliative radiotherapy will be allowed as described in the Prior and Concomitant Therapy section)
  * Radiotherapy during study or within 4 weeks of start of study drug. (Palliative radiotherapy will be allowed as described in the Prior and Concomitant Therapy section) (FOR FRANCE ONLY)
  * Major surgery, open biopsy or significant traumatic injury within 4 weeks of first dose of study drug (bronchoscopy is allowed)
  * Granulocyte colony stimulating factor (GCSF) or Granulocyte macrophage colony stimulating factor (GMCSF), within 3 weeks of study entry (these growth factors may be used during the study thereafter).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 904 (Actual)
Dates: Start 2007-02; Primary Completion 2010-04 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (105):
- Austria (3):
  - Innsbruck
  - Linz
  - Vienna
- Belgium (6):
  - Brasschaat
  - Bruxelles - Brussel
  - Edegem
  - Leuven
  - Liège
  - Namur
- Brazil (10):
  - Salvador, Estado de Bahia
  - Brasília, Federal District
  - Goiânia, Goiás
  - Belo Horizonte, Minas Gerais
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - Jaú, São Paulo
  - Santo André, São Paulo
  - São Paulo, São Paulo
  - Sorocaba, São Paulo
- Montreal, Quebec, Canada
- China (6):
  - Guangzhou, Guangdong
  - Wuhan, Hubei
  - Nanjing, Jiangsu
  - Hangzhou, Zhejiang
  - Beijing
  - Shanghai
- Nicosia, Cyprus
- Finland (3):
  - HUS
  - Preitilä
  - Tampere
- France (12):
  - Bayonne
  - Grenoble
  - Hyères
  - Le Mans
  - Marseille
  - Nantes
  - Nîmes
  - Paris
  - Perpignan
  - Pierre-Bénite
  - Strasbourg
  - Tours
- Germany (12):
  - Heidelberg, Baden-Wurttemberg
  - Karlsruhe, Baden-Wurttemberg
  - Löwenstein, Baden-Wurttemberg
  - Gauting, Bavaria
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Hofheim, Hesse
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Leipzig, Saxony
  - Großhansdorf, Schleswig-Holstein
  - Bad Berka, Thuringia
- Greece (3):
  - Heraklion, Crete
  - Athens, Greece
  - Athens
- Hungary (5):
  - Budapest
  - Deszk
  - Mátraháza
  - Székesfehérvár
  - Törökbálint
- Israel (5):
  - Ashkelon
  - Holon
  - Kfar Saba
  - Rehovot
  - Tel Litwinsky
- Italy (12):
  - Rozzano, Milano
  - Monza, Monza-Brianza
  - Aviano, Pordenone
  - Bologna
  - Catania
  - Florence
  - Livorno
  - Milan
  - Roma
  - Sassari
  - Venezia
  - Verona
- Mexico (3):
  - Guadalajara, Jalisco
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
- Netherlands (5):
  - 's-Hertogenbosch
  - Ede
  - Harderwijk
  - Heerlen
  - Nieuwegein
- Spain (8):
  - A Coruña, A Coruña
  - Barcelona, Barcelona
  - Terrassa, Barcelona
  - Cruces/Barakaldo, Bilbao
  - Madrid, Madrid
  - Málaga, Málaga
  - Seville, Sevilla
  - Valencia, Valencia
- Switzerland (3):
  - Basel, Canton of Basel-City
  - Bern, Canton of Bern
  - Genéve, Canton of Geneva
- United Kingdom (7):
  - Cambridge, Cambridgeshire
  - Aberdeen, Grampian
  - Leicester, Leicestershire
  - London, London
  - Sutton, Surrey
  - Wolverhampton, West Midlands
  - Birmingham

REFERENCES:
- [Result] Paz-Ares LG, Biesma B, Heigener D, von Pawel J, Eisen T, Bennouna J, Zhang L, Liao M, Sun Y, Gans S, Syrigos K, Le Marie E, Gottfried M, Vansteenkiste J, Alberola V, Strauss UP, Montegriffo E, Ong TJ, Santoro A; NSCLC [non-small-cell lung cancer] Research Experience Utilizing Sorafenib (NExUS) Investigators Study Group. Phase III, randomized, double-blind, placebo-controlled trial of gemcitabine/cisplatin alone or with sorafenib for the first-line treatment of advanced, nonsquamous non-small-cell lung cancer. J Clin Oncol. 2012 Sep 1;30(25):3084-92. doi: 10.1200/JCO.2011.39.7646. Epub 2012 Jul 30. PMID 22851564
- See also: Click here and search for Bayer Product information provided by EMA — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 93 centers across 16 countries, which enrolled and randomized at least one patient. From a total of 1011 patients who were screened, 904 patients were randomized between 23 FEB 2007 and 03 MAR 2009.
Pre-assignment Details: All 904 randomized patients were included in the intent to treat (ITT) population. A total of 901 patients received at least one dose of study medication and were included in the safety population. Study medication included administration of any one of the following treatments: gemcitabine, cisplatin, sorafenib or placebo.
Period: Treatment Period
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Started | 452 | 452 (Reasons for not treated: Adverse event (N=1); Consent withdrawn (N=1); Reason missing (N=1))
Received Treatment | 452 | 449
Completed | 0 | 0
Not Completed | 452 | 452
Not completed — Adverse Event | 117 | 83
Not completed — Death | 21 | 12
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 4 | 5
Not completed — Protocol Violation | 8 | 7
Not completed — Disease Progression | 231 | 288
Not completed — Consent Withdrawn | 36 | 20
Not completed — Amended Protocol Criteria | 22 | 18
Not completed — Non-compliance | 7 | 8
Not completed — Second Malignancy | 0 | 1
Not completed — Reason Missing | 0 | 4
Not completed — Treatment Ongoing | 6 | 4
Period: Follow-up Period
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Started | 425 (425 entered, comprising 452 randomized less 21 deaths & 6 ongoing on treatment) | 434 (434 entered, comprising 452 randomized less 12 deaths, 2 lost to follow-up & 4 ongoing on treatment)
Completed | 0 | 0
Not Completed | 425 | 434
Not completed — Death | 299 | 311
Not completed — Lost to Follow-up | 6 | 10
Not completed — Reason Missing | 120 | 113

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC | Total
Number analyzed (Participants) | 452 | 452 | 904
Age, Continuous [Median (Full Range); unit: Years] | 60 [28 to 81] | 59 [22 to 82] | 59 [22 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 155 | 323
  Male | 284 | 297 | 581
histology of the tumor [Number; unit: Participants]
  Non-squamous | 385 | 387 | 772
  Squamous | 67 | 65 | 132
Time since initial diagnosis [Median (Full Range); unit: Weeks] | 2.6 [0 to 552] | 2.9 [0 to 924] | 2.7 [0 to 924]
Smoking history [Number; unit: Participants]
  Non-smoker | 111 | 107 | 218
  Passive smoker | 2 | 3 | 5
  Past or present smoker | 338 | 342 | 680
  Not available | 1 | 0 | 1
Tumor stage at randomization [Number; unit: Participants] — Categorized information on tumor size, lymph node involvement and metastases. Stages I-IV. The higher the stage the more advanced cancer. Stage IIIB versus IV was a stratification factor for randomization. Stage IIIB (according to American Joint Committee on Cancer): primary tumor any stage, regional lymph node stage N3, no distant metastasis OR primary tumor stage T4, regional lymph node any stage, no distant metastasis. Stage IV: primary tumor any stage, regional lymph node any stage, distant metastasis present.
  Participants
    Stage III B | 57 | 55 | 112
    Stage IV | 395 | 397 | 792
ECOG (Eastern Cooperative Oncology Group) Performance Status at randomization [Number; unit: Participants] — ECOG 0 versus 1 was a stratification factor for randomization. ECOG Performance Status is a rating of daily living abilities, from 0 to 5: 0= fully active without restriction. 1= restricted in physically strenuous activity; 2= ambulatory, capable of all selfcare; 3= capable of limited selfcare; 4= completely disabled; 5= dead.
  Participants
    0 | 176 | 175 | 351
    1 | 276 | 277 | 553

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in the ITT (Non-squamous) Population
Description: Overall survival (OS) was defined as the time from date of randomization to death due to any cause. Patients still alive at the time of analysis were censored at their last date of last contact.
Time Frame: from randomization of the first patient until 38 months or date of death of any cause whichever came first
Population: Evaluation of OS based on ITT (non-squamous) population. Patients alive at the time of analysis were censored at their last date of follow-up (last visit or contact or at the data cut-off date). In the case of an incomplete date, where day was missing, day 15 (the middle of the month) was used.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Number analyzed (Participants) | 385 | 387
days | 376 [333 to 416] | 379 [335 to 414]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + GC vs Placebo + GC; Sample size based on the primary efficacy endpoint of OS in the ITT (non-squamous) population. Clinically meaningful improvement defined as 30% increase in median OS (that is, a hazard ratio of 0.76923, Sorafenib+GC over Placebo+GC). With one-sided alpha of 0.025, power of 86% and a randomization ratio of 1:1 between Sorafenib+GC and Placebo+GC, and one formal final analysis of OS performed, a total of 544 events (deaths) were required; Test type: Superiority or Other; p = 0.401, Log Rank; Two treatment groups compared using a log-rank test with one-sided alpha of 0.025 stratified by the same stratification factors as randomization; Hazard Ratio (HR) = 0.98, 95% CI [0.83 to 1.16]

2. Secondary Outcome: OS in the ITT (Both Squamous and Non-squamous) Population
Description: OS was defined as the time from date of randomization to death due to any cause. Patients still alive at the time of analysis were censored at their last date of last contact.
Time Frame: from randomization of the first patient until 38 months or date of death of any cause whichever came first
Population: Evaluation of OS based on ITT (both non-squamous and squamous) population. Patients alive at the time of analysis were censored at their last date of follow-up (last visit or contact or at the data cut-off date). In the case of an incomplete date, where day was missing, day 15 (the middle of the month) was used.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Number analyzed (Participants) | 452 | 452
days | 371 [322 to 410] | 378 [335 to 412]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + GC vs Placebo + GC; Test type: Superiority or Other; p = 0.563, Log Rank; Two treatment groups compared using a log-rank test with one-sided alpha of 0.025 stratified by the same factors as randomization plus histology; Hazard Ratio (HR) = 1.01, 95% CI [0.87 to 1.18]

3. Secondary Outcome: OS in the ITT (Squamous) Population
Description: as for outcome 2
Time Frame: from randomization of the first patient until 38 months or date of death of any cause whichever came first
Population: Evaluation of OS based on ITT (squamous) population. Patients alive at the time of analysis were censored at their last date of follow-up (last visit or contact or at the data cut-off date). In the case of an incomplete date, where day was missing, day 15 (the middle of the month) was used. No statistical testing performed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Number analyzed (Participants) | 67 | 65
days | 254 [197 to 455] | 374 [282 to 519]

4. Secondary Outcome: Progression-free Survival (PFS) in the ITT (Non-squamous) Population
Description: PFS was defined as the time from date of randomization to disease progression (radiological or clinical, whichever was earlier, based on Investigator-assessment using Response Evaluation Criteria in Solid Tumors (RECIST), version 1.0) or death due to any cause, whichever occured first. Patients without progression or death at the time of analysis were censored at their last date of tumor evaluation. Disease progression: increase in the sum of tumor lesion sizes or new lesions.
Time Frame: from randomization of the first patient until 38 months or date of death or progression whichever came first, assessed until discontinuation every 6 weeks up to 9 months and then every 12 weeks
Population: Evaluation of PFS based on ITT (non-squamous) population. PFS for patients with no tumour assessments after baseline was censored at one day.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Number analyzed (Participants) | 385 | 387
days | 183 [168 to 208] | 168 [156 to 174]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + GC vs Placebo + GC; Test type: Superiority or Other; p = 0.008, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.83, 95% CI [0.71 to 0.97]

5. Secondary Outcome: Time to Progression (TTP) in the ITT (Non-squamous) Population
Description: TTP was defined as the time from date of randomization to disease progression (radiological or clinical, whichever was earlier, based on Investigator-assessment using RECIST version 1.0). Patients without progression at the time of analysis or death before progression were censored at their last date of tumor evaluation. Disease progression: increase in the sum of tumor lesion sizes or new lesions.
Time Frame: as for outcome 4
Population: Evaluation of TTP based on ITT (non-squamous) population. TTP for patients with no tumour assessments after baseline was censored at one day.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Number analyzed (Participants) | 385 | 387
days | 185 [171 to 210] | 167 [156 to 173]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + GC vs Placebo + GC; Test type: Superiority or Other; p = 0.0004, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.73, 95% CI [0.60 to 0.88]

6. Secondary Outcome: Percentage of Participants With Different Tumor Response in the ITT (Non-squamous) Population
Description: Tumor response (= Best Overall Response) of a patient was defined as the best tumor response (confirmed Complete Response (CR: disappearance of tumor lesions), confirmed Partial Response (PR: a decrease of at least 30% in the sum of tumor lesion sizes), Stable Disease (SD: steady state of disease), or Progressive Disease (PD: an increase in the sum of tumor lesions sizes or new lesions)) observed during trial period assessed according to the RECIST criteria (version 1.0) based on Investigator-assessment.
Time Frame: as for outcome 4
Population: Evaluation of Tumour Response based on ITT (non-squamous) population.
Measure: Number; unit: percentage of participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Number analyzed (Participants) | 385 | 387
percentage of participants
  CR | 0.0 [0.0 to 0.8] | 0.0 [0.0 to 0.8]
  confirmed PR | 27.8 [23.4 to 32.6] | 25.8 [21.6 to 30.5]
  SD | 34.3 [29.6 to 39.3] | 37.2 [32.4 to 42.2]
  PD | 10.9 [8.0 to 14.5] | 17.1 [13.4 to 21.2]
  Not assessable | 27.0 [22.6 to 31.7] | 19.9 [16.0 to 24.2]
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + GC vs Placebo + GC; Test type: Superiority or Other; p = 0.2733, Cochran-Mantel-Haenszel; Two treatment groups compared using a CMH test with one-sided alpha of 0.025 stratified by the same stratification factors as randomization; Difference in Tumour Response (CR+PR) = -1.92, 95% CI [-8.19 to 4.34]

7. Secondary Outcome: Disease Control (DC) in the ITT (Non-squamous) Population
Description: DC was defined as the total number of patients whose best response was not PD according to RECIST (version 1.0) by Investigator-assessment (= total number of CR + total number of PR + total number of SD; CR or PR had to be maintained for at least 28 days from the first demonstration of that rating, SD had to be documented at least once more than 6 weeks from baseline). PD: an increase in the sum of tumor lesions sizes or new lesions.
Time Frame: as for outcome 4
Population: Evaluation of Disease Control based on ITT (non-squamous) population.
Measure: Number; unit: percentage of participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Number analyzed (Participants) | 385 | 387
percentage of participants | 62.1 | 63.1
Statistical Analysis 1: Comparison: Sorafenib (Nexavar, BAY43-9006) + GC vs Placebo + GC; Test type: Superiority or Other; p = 0.3902, Cochran-Mantel-Haenszel; [statistical method as in outcome 6, analysis 1]; Difference in Disease Control = 0.97, 95% CI [-5.87 to 7.81]

8. Secondary Outcome: Duration of Response in the ITT (Non-squamous) Population
Description: Duration of response was defined as the time from date of first documented objective response of PR or CR, whichever was noted earlier, to date of disease progression or death (if death occurred before progression was documented). Patients without disease progression at the time of analysis or death before progression were censored at the last date of tumor evaluation. Disease progression: increase in the sum of tumor lesion sizes or new lesions.
Time Frame: as for outcome 4
Population: Evaluation of duration of response based on ITT (non-squamous) population. No statistical testing performed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Number analyzed (Participants) | 107 | 100
days | 171 [147 to 203] | 133 [126 to 146]

9. Secondary Outcome: Duration of Stable Disease (SD) in the ITT (Non-squamous) Population
Description: Duration of SD was defined as the time from date of randomization to date that disease progression (radiological or clinical, whichever was earlier) was first documented. Patients without disease progression at the time of analysis or death before progression were censored at the date of their last tumor assessment.(Disease progression: increase in the sum of tumor lesion sizes or new lesions.) Duration of stable disease was only evaluated in patients failing to achieve a best response of CR or PR.
Time Frame: as for outcome 4
Population: Evaluation of duration of stable disease based on ITT (non-squamous) population. No statistical testing performed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Number analyzed (Participants) | 174 | 210
days | 144 [126 to 168] | 131 [125 to 156]

10. Secondary Outcome: Time to Response (TTR) in the ITT (Non-squamous) Population
Description: TTR for patients who achieved a best response (CR or PR) was defined as the time from date of randomization to the earliest date that response was first documented.
Time Frame: from randomization of the first patient until 38 months or date of death of any cause whichever came first
Population: Evaluation of TTR based on ITT (non-squamous) population. No statistical testing performed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Number analyzed (Participants) | 107 | 100
days | 42 [41 to 44] | 43 [42 to 44]

11. Secondary Outcome: Functional Assessment of Cancer Treatment-Lung (FACT-L) Scores in the ITT (Non-squamous) Population
Description: The FACT-L measures health related quality of life (HRQOL) and composes of five domains: the four domains (physical well being, emotional well being, social well being, functional well being) from the Functional Assessment of Cancer Treatment-General scale (FACT-G) and the lung cancer subscale (LCS). The FACT-L total score ranges from 0 to 136, higher scores represent better HRQOL.
Time Frame: from randomization of the first patient until 38 months
Population: All patients valid for the ITT analysis who have a baseline and at least one post baseline value.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Number analyzed (Participants) | 282 | 283
scores on a scale
  cycle 2 (day 22) | 90.6 [88.5 to 92.6] | 94.0 [92.2 to 95.9]
  cycle 4 (day 64) | 90.1 [88.1 to 92.2] | 93.6 [91.7 to 95.4]
  cycle 6 (day 106) | 89.7 [87.5 to 91.8] | 93.1 [91.1 to 95.1]

12. Secondary Outcome: Lung Cancer Subscale (LCS) Scores in the ITT (Non-squamous) Population
Description: LCS is a subscale of FACT-L measuring lung cancer specific symptoms. The LCS scores range from 0 to 28, higher scores represent fewer lung cancer symptoms.
Time Frame: from randomization of the first patient to 38 months later or death whatever occurs first.
Population: All patients valid for the ITT analysis who have a baseline and at least one post baseline value.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Number analyzed (Participants) | 314 | 317
scores on a scale
  cycle 1 (day 1) | 20.0 [19.6 to 20.4] | 20.5 [20.1 to 20.9]
  cycle 2 (day 22) | 19.9 [19.5 to 20.4] | 20.5 [20.1 to 20.8]
  cycle 3 (day 43) | 19.9 [19.4 to 20.3] | 20.4 [20.0 to 20.8]
  cycle 4 (day 64) | 19.8 [19.4 to 20.2] | 20.3 [19.9 to 20.7]
  cycle 5 (day 85) | 19.7 [19.3 to 20.2] | 20.3 [19.8 to 20.7]
  cycle 6 (day 106) | 19.7 [19.2 to 20.1] | 20.2 [19.7 to 20.6]

13. Secondary Outcome: Time to Symptomatic Deterioration (TSD) in the ITT (Non-squamous) Population
Description: TSD is defined as the time from randomization to the date of symptomatic deterioration (≥3 point decline in the LCS score that is maintained for at least 2 consecutive cycles) or death if death occurs before these 2 consecutive cycles are completed.
Time Frame: from randomization of the first patient to 38 months later or death whatever occurs first
Population: All patients valid for the ITT analysis who have a baseline and at least one post baseline value.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Number analyzed (Participants) | 321 | 333
months | 6.9 [5.8 to 8.7] | 4.5 [3.6 to 5.9]

14. Secondary Outcome: Euro Quality of Life - 5D (EQ-5D) Index Scores in the ITT (Non-squamous) Population
Description: The EQ-5D contains a descriptive system which measures 5 health dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. These five health dimensions are summarized into a single score, the EQ-5D index score which ranges from -0.594 to 1 when the United Kingdom (UK) weights are applied (0=death, 1=perfect health). Higher index scores represent better health states.
Time Frame: from randomization of the first patient until 38 months later or death whatever occurs first
Population: All patients valid for the ITT analysis who have a baseline and at least one post baseline value.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Number analyzed (Participants) | 323 | 318
scores on a scale
  cycle 1 (day 1) | 0.70 [0.67 to 0.72] | 0.76 [0.73 to 0.78]
  cycle 2 (day 22) | 0.69 [0.67 to 0.72] | 0.75 [0.73 to 0.78]
  cycle 3 (day 43) | 0.69 [0.66 to 0.71] | 0.75 [0.72 to 0.77]
  cycle 4 (day 64) | 0.68 [0.66 to 0.71] | 0.74 [0.72 to 0.76]
  cycle 5 (day 85) | 0.68 [0.65 to 0.70] | 0.73 [0.71 to 0.76]
  cycle 6 (day 106) | 0.67 [0.64 to 0.70] | 0.73 [0.70 to 0.75]

15. Secondary Outcome: EQ-5D Visual Analog Scale (VAS) Scores in the ITT (Non-squamous) Population
Description: The EQ-5D also contains a visual analog scale (EQ-VAS), which records the respondent's self-rated health status on a vertical graduated visual analog scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: from randomization of the first patient until 38 months later or death whatever occurs first
Population: All patients valid for the ITT analysis who have a baseline and at least one post baseline value.
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Number analyzed (Participants) | 315 | 313
scores on a scale
  cycle 1 (day 1) | 66.43 [64.65 to 68.21] | 68.96 [67.18 to 70.73]
  cycle 2 (day 22) | 66.43 [64.68 to 68.18] | 68.96 [67.19 to 70.72]
  cycle 3 (day 43) | 66.43 [64.68 to 68.18] | 68.95 [67.18 to 70.72]
  cycle 4 (day 64) | 66.43 [64.65 to 68.20] | 68.95 [67.15 to 70.75]
  cycle 5 (day 85) | 66.42 [64.61 to 68.24] | 68.95 [67.10 to 70.80]
  cycle 6 (day 106) | 66.42 [64.55 to 68.30] | 68.95 [67.02 to 70.87]

ADVERSE EVENTS:
Description: Acronyms used: Absolute Neutrophil Count (ANC), Central Nervous System (CNS), Gastro-Intestinal (GI), Glomerular Filtration Rate (GFR), International Normalized Ratio (INR), Not Otherwise Specified (NOS), Alanine transaminase (ALT), Aspartate transaminase (AST), Acute respiratory distress syndrome (ARDS), cranial nerve (CN)
Arm/Group | Sorafenib (Nexavar, BAY43-9006) + GC | Placebo + GC
Serious Adverse Events (participants affected / at risk) | 270/452 | 198/449
Other Adverse Events (participants affected / at risk) | 440/452 | 435/449
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) + GC (N=452) | Placebo + GC (N=449)
Blood - Other (Blood and lymphatic system disorders) | 3 | 2
Bone marrow cellularity (Blood and lymphatic system disorders) | 1 | 0
Edema: Head and Neck (Blood and lymphatic system disorders) | 0 | 1
Edema: Limb (Blood and lymphatic system disorders) | 3 | 1
Hemoglobin (Blood and lymphatic system disorders) | 18 | 12
INR (Blood and lymphatic system disorders) | 1 | 0
Leukocytes (Blood and lymphatic system disorders) | 12 | 5
Neutrophils (Blood and lymphatic system disorders) | 19 | 12
Platelets (Blood and lymphatic system disorders) | 63 | 27
Cardiac arrhythmia - Other (Cardiac disorders) | 1 | 0
Cardiac general - Other (Cardiac disorders) | 1 | 1
Cardiac ischemia/infarction (Cardiac disorders) | 9 | 9
Cardiopulmonary arrest (Cardiac disorders) | 1 | 1
Conduction abnormality, Conduction abnormality NOS (Cardiac disorders) | 0 | 1
Hypertension (Cardiac disorders) | 3 | 1
Hypotension (Cardiac disorders) | 4 | 2
Left ventricular systolic dysfunction (Cardiac disorders) | 2 | 1
Pericardial effusion (Cardiac disorders) | 4 | 5
Pericarditis (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia, Atrial fibrillation (Cardiac disorders) | 6 | 1
Supraventricular arrhythmia, Atrial flutter (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia, Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Ventricular arrhythmia, Ventricular arrhythmia NOS (Cardiac disorders) | 0 | 1
Ventricular arrhythmia, Ventricular tachycardia (Cardiac disorders) | 2 | 0
Diabetes (Endocrine disorders) | 1 | 0
Endocrine - Other (Endocrine disorders) | 0 | 1
Optic disc edema (Eye disorders) | 0 | 1
Vitreous hemorrhage (Eye disorders) | 1 | 0
Anorexia (Gastrointestinal disorders) | 6 | 0
Ascites (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 3
Dehydration (Gastrointestinal disorders) | 0 | 4
Diarrhea (Gastrointestinal disorders) | 7 | 2
Dysphagia (Gastrointestinal disorders) | 3 | 2
Enteritis (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 3 | 0
GI - Other (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Mucositis (functional/symptomatic), Esophagus (Gastrointestinal disorders) | 1 | 0
Mucositis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 14 | 6
Obstruction, GI, Colon (Gastrointestinal disorders) | 1 | 3
Obstruction, GI, Gallbladder (Gastrointestinal disorders) | 1 | 0
Obstruction, GI, Ileum (Gastrointestinal disorders) | 0 | 1
Perforation, GI, Colon (Gastrointestinal disorders) | 1 | 0
Perforation, GI, Stomach (Gastrointestinal disorders) | 1 | 0
Stricture, GI, Colon (Gastrointestinal disorders) | 0 | 2
Stricture, GI, Esophagus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 10 | 11
Constitutional symptoms - Other (General disorders) | 11 | 2
Death not associated with CTCAE term, Death NOS (General disorders) | 1 | 4
Death not associated with CTCAE term, Disease progression NOS (General disorders) | 21 | 15
Death not associated with CTCAE term, Multi-Organ Failure (General disorders) | 2 | 5
Death not associated with CTCAE term, Sudden death (General disorders) | 0 | 1
Fatigue (General disorders) | 11 | 4
Fever (General disorders) | 14 | 6
Hypothermia (General disorders) | 0 | 1
No code in CTCAE (General disorders) | 1 | 1
Pain, Abdomen NOS (General disorders) | 8 | 3
Pain, Back (General disorders) | 3 | 3
Pain, Bone (General disorders) | 4 | 2
Pain, Chest wall (General disorders) | 1 | 1
Pain, Chest/Thorax NOS (General disorders) | 3 | 1
Pain, Extremity - limb (General disorders) | 0 | 1
Pain, Gallbladder (General disorders) | 1 | 0
Pain, Head/Headache (General disorders) | 2 | 0
Pain, Neuralgia/Peripheral nerve (General disorders) | 0 | 1
Pain, Other (General disorders) | 2 | 0
Pain, Pelvis (General disorders) | 1 | 0
Pain, Stomach (General disorders) | 1 | 0
Pain, Tumor pain (General disorders) | 2 | 1
Tumor lysis syndrome (General disorders) | 1 | 0
Weight loss (General disorders) | 1 | 0
Hepatobiliary - Other (Hepatobiliary disorders) | 3 | 0
Liver dysfunction (Hepatobiliary disorders) | 0 | 1
Pancreatitis (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 0
Febrile neutropenia (Infections and infestations) | 10 | 6
Infection (Documented clinically), Bladder (urinary) (Infections and infestations) | 1 | 0
Infection (Documented clinically), Blood (Infections and infestations) | 3 | 0
Infection (Documented clinically), Bronchus (Infections and infestations) | 0 | 1
Infection (Documented clinically), Kidney (Infections and infestations) | 1 | 0
Infection (Documented clinically), Lung (Pneumonia) (Infections and infestations) | 4 | 4
Infection (Documented clinically), Pleura (Empyema) (Infections and infestations) | 0 | 1
Infection (Documented clinically), Upper airway NOS (Infections and infestations) | 1 | 0
Infection - Other (Infections and infestations) | 2 | 1
Infection with normal ANC, Abdomen NOS (Infections and infestations) | 1 | 1
Infection with normal ANC, Anal/perianal (Infections and infestations) | 1 | 0
Infection with normal ANC, Blood (Infections and infestations) | 1 | 0
Infection with normal ANC, Bronchus (Infections and infestations) | 6 | 3
Infection with normal ANC, Catheter-related (Infections and infestations) | 1 | 0
Infection with normal ANC, Lung (Pneumonia) (Infections and infestations) | 22 | 11
Infection with normal ANC, Meninges (Meningitis) (Infections and infestations) | 1 | 0
Infection with normal ANC, Scrotum (Infections and infestations) | 0 | 1
Infection with normal ANC, Skin (cellulitis) (Infections and infestations) | 1 | 0
Infection with normal ANC, Soft tissue NOS (Infections and infestations) | 1 | 0
Infection with normal ANC, Urinary tract NOS (Infections and infestations) | 1 | 0
Infection with unknown ANC, Blood (Infections and infestations) | 1 | 1
Infection with unknown ANC, Lung (Pneumonia) (Infections and infestations) | 6 | 2
Infection with unknown ANC, Pleura (Empyema) (Infections and infestations) | 2 | 0
Infection with unknown ANC, Soft tissue NOS (Infections and infestations) | 1 | 0
Infection with unknown ANC, Wound (Infections and infestations) | 1 | 0
Intraop injury, Jejunum (Injury, poisoning and procedural complications) | 1 | 0
Intraop injury, Lung (Injury, poisoning and procedural complications) | 1 | 2
ALT (Metabolism and nutrition disorders) | 1 | 0
Bilirubin (Hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 | 0
Creatinine (Metabolism and nutrition disorders) | 4 | 2
GFR (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 0
Hyponatremia (Metabolism and nutrition disorders) | 6 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 4
Muscle weakness, Extremity - lower (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness, Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue necrosis, Extremity - lower (Musculoskeletal and connective tissue disorders) | 0 | 1
CNS ischemia (Nervous system disorders) | 6 | 3
Confusion (Nervous system disorders) | 1 | 2
Mood alteration, Depression (Nervous system disorders) | 0 | 1
Neurology - Other (Nervous system disorders) | 1 | 2
Neuropathy: Cranial, CN II Vision (Nervous system disorders) | 0 | 1
Neuropathy: motor (Nervous system disorders) | 1 | 0
Neuropathy: sensory (Nervous system disorders) | 0 | 1
Personality (Nervous system disorders) | 1 | 0
Pyramidal tract dysfunction (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 4 | 3
Somnolence (Nervous system disorders) | 2 | 1
Speech impairment (Nervous system disorders) | 0 | 2
Syncope (Fainting) (Nervous system disorders) | 3 | 2
Tremor (Nervous system disorders) | 1 | 0
Renal - Other (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 4 | 2
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Airway obstruction, Bronchus (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 23 | 26
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dermatology - Other (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 0
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 | 1
Artery injury, Aorta (Vascular disorders) | 1 | 0
CNS hemorrhage (Vascular disorders) | 2 | 3
Hemorrhage - Other (Vascular disorders) | 2 | 0
Hemorrhage pulmonary, Bronchopulmonary NOS (Vascular disorders) | 5 | 1
Hemorrhage pulmonary, Lung (Vascular disorders) | 5 | 2
Hemorrhage pulmonary, Nose (Vascular disorders) | 3 | 2
Hemorrhage pulmonary, Respiratory tract NOS (Vascular disorders) | 1 | 0
Hemorrhage, GI, Abdomen NOS (Vascular disorders) | 1 | 0
Hemorrhage, GI, Anus (Vascular disorders) | 3 | 1
Hemorrhage, GI, Colon (Vascular disorders) | 1 | 0
Hemorrhage, GI, Duodenum (Vascular disorders) | 1 | 0
Hemorrhage, GI, Rectum (Vascular disorders) | 1 | 0
Hemorrhage, GI, Stomach (Vascular disorders) | 2 | 1
Hemorrhage, GI, Upper GI NOS (Vascular disorders) | 1 | 1
Peripheral arterial ischemia (Vascular disorders) | 4 | 4
Phlebitis (Vascular disorders) | 0 | 3
Thrombosis/Embolism (vascular access) (Vascular disorders) | 3 | 5
Thrombosis/Thrombus/Embolism (Vascular disorders) | 26 | 22
Vascular - Other (Vascular disorders) | 1 | 2
Visceral arterial ischemia (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) + GC (N=452) | Placebo + GC (N=449)
Blood - Other (Blood and lymphatic system disorders) | 16 | 34
Edema: Limb (Blood and lymphatic system disorders) | 22 | 39
Hemoglobin (Blood and lymphatic system disorders) | 214 | 221
Leukocytes (Blood and lymphatic system disorders) | 158 | 146
Lymphopenia (Blood and lymphatic system disorders) | 30 | 17
Neutrophils (Blood and lymphatic system disorders) | 210 | 225
Platelets (Blood and lymphatic system disorders) | 255 | 210
Hypertension (Cardiac disorders) | 76 | 34
Tinnitus (Ear and labyrinth disorders) | 24 | 34
Anorexia (Gastrointestinal disorders) | 177 | 158
Constipation (Gastrointestinal disorders) | 148 | 133
Diarrhea (Gastrointestinal disorders) | 189 | 80
Dysphagia (Gastrointestinal disorders) | 26 | 8
Heartburn (Gastrointestinal disorders) | 37 | 32
Mucositis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 114 | 50
Nausea (Gastrointestinal disorders) | 263 | 247
Taste Alteration (Gastrointestinal disorders) | 27 | 32
Vomiting (Gastrointestinal disorders) | 199 | 198
Fatigue (General disorders) | 242 | 237
Fever (General disorders) | 67 | 59
Insomnia (General disorders) | 51 | 55
Pain, Abdomen NOS (General disorders) | 61 | 42
Pain, Back (General disorders) | 46 | 37
Pain, Chest/Thorax NOS (General disorders) | 54 | 64
Pain, Extremity - limb (General disorders) | 32 | 35
Pain, Head/Headache (General disorders) | 54 | 43
Pain, Joint (General disorders) | 24 | 25
Pain, Muscle (General disorders) | 24 | 18
Pain, Stomach (General disorders) | 27 | 28
Pain, Throat/Pharynx/Larynx (General disorders) | 23 | 10
Weight loss (General disorders) | 55 | 31
Infection with normal ANC, Upper airway NOS (Infections and infestations) | 26 | 27
ALT (Metabolism and nutrition disorders) | 27 | 24
AST (Metabolism and nutrition disorders) | 25 | 12
Creatinine (Metabolism and nutrition disorders) | 27 | 39
Hypocalcemia (Metabolism and nutrition disorders) | 49 | 20
Hypokalemia (Metabolism and nutrition disorders) | 75 | 43
Hypomagnesemia (Metabolism and nutrition disorders) | 67 | 55
Hyponatremia (Metabolism and nutrition disorders) | 49 | 44
Hypophosphatemia (Metabolism and nutrition disorders) | 31 | 12
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 37 | 44
Dizziness (Nervous system disorders) | 55 | 46
Neuropathy: sensory (Nervous system disorders) | 71 | 77
Cough (Respiratory, thoracic and mediastinal disorders) | 80 | 106
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 92 | 86
Voice changes (Respiratory, thoracic and mediastinal disorders) | 34 | 23
Alopecia (Skin and subcutaneous tissue disorders) | 148 | 74
Dermatology - Other (Skin and subcutaneous tissue disorders) | 25 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 32 | 15
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 121 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 36 | 19
Rash/desquamation (Skin and subcutaneous tissue disorders) | 165 | 93
Hemorrhage pulmonary, Nose (Vascular disorders) | 78 | 33

LIMITATIONS AND CAVEATS:
Inclusion of squamous patients stopped in FEB 2008, as 11961 (NCT00558636) trial reported higher mortality for this subgroup. Squamous patients in 12006 (NCT00449033) trial discontinued drug as a precaution endorsed by Data Monitoring Committee.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator, whilst free to use data from the study for scientific purposes, must not publish any document relating to the Trial without first notifying Bayer in writing and obtaining written consent. Bayer recognizes the right of the investigator to publish the results upon completion of the study. The investigator must send a draft manuscript of the publication or abstract to Bayer 60 days ahead of submission to obtain approval prior to submission of the final version for publication.